CLINICAL TRIAL: NCT00502229
Title: What is the Following Step to Improve Fertility in Infertile PCOS Patients Ovulating Under Clomiphene Citrate or Metformin? A Randomized Controlled Clinical Study.
Brief Title: Therapy for Infertile PCOS Patients Ovulating Under Clomiphene Citrate or Metformin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05/2006c
Record Dates: First submitted 2007-07-12; First posted 2007-07-17 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Polycystic Ovary Syndrome; Infertility
Keywords: Clomiphene citrate; Controlled overian stimulation; Infertility; Metformin; Polycystic ovary syndrome; Treatment
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Clomiphene; Metformin

ARMS (2):
- Group A (Active Comparator): Continuing treatment
  Interventions: Drug: Clomiphene citrate, metformin, highly purified urinary FSH
- Group B (Active Comparator): Gonadotrophins
  Interventions: Drug: Clomiphene citrate, metformin, highly purified urinary FSH

INTERVENTIONS:
Drug: Clomiphene citrate, metformin, highly purified urinary FSH

SUMMARY:
Several data demonstrated that both clomiphene citrate (CC) and metformin are two safe and valid first-step options to induce ovulation in infertile anovulatory PCOS patients. Notwithstanding a high percentage of patients ovulate under treatment, only ~40% and 60% of subjects obtain a pregnancy after CC and metformin, respectively.

For these patients, controlled ovarian stimulation (COS) followed by intrauterine insemination (IUI) could be the next therapeutic step before assisted reproductive techniques since IUI improves significantly the fertility in couples with unexplained infertility. Furthermore, to date it is not defined if COS should be obtained using the same ovulatory agent (CC or metformin) or switching the treatment to gonadotropins.

In this view, the aim of the present study will be to evaluate the best management of infertile PCOS patients ovulating after CC or metformin.

DETAILED DESCRIPTION:
Infertile PCOS patients who ovulated under CC or metformin without pregnancy achievement will be enrolled and treated with three trials of COS plus IUI. All patients will be randomly allocated into two different groups (groups A and B). In group A, COS will be obtained using the same ovulatory agent (CC or metformin) employed in the previous ovulatory cycles, whereas in group B using gonadotropins in a low-dose step-up regimen.

All patients eligible will undergo baseline assessment consisting of anthropometric, hormonal, and ultrasonographic evaluations. During the study, the clinical and reproductive outcomes, and the adverse experience will be evaluated and the will be analyzed also categorizing the patients according to ovulatory agent used for COS (CC or metformin).

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant. Continuous variables will be analyzed with the unpaired t test and general linear model for repeated measures analysis with Bonferroni test for the post-hoc analysis as required. For categorical variables, the Pearson chi-square and Fisher's exact tests will be used. Cumulative pregnancy rate, our primary end-point, will be calculated by the Kaplan-Maier method, and the differences between the two groups will be assessed with the log-rank test. Cox proportional-hazards model will be used to calculate the hazard ratio for new pregnancy in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Polycystic ovary syndrome (using NIH criteria)
* Anovulatory infertility (using WHO criteria)

Exclusion Criteria:

* Age <18 or >35 years
* Severe obesity (BMI >35)
* Neoplastic, metabolic, hepatic, and cardiovascular disorders or other concurrent medical illnesses
* Hypothyroidism, hyperprolactinemia, Cushing's syndrome, and non-classical congenital adrenal hyperplasia
* Current or previous (within the last six months) use of oral contraceptives, glucocorticoids, antiandrogens, antidiabetic and anti-obesity drugs or other hormonal drugs
* Intention to start a diet or a specific program of physical activity
* Organic pelvic diseases
* Previous pelvic surgery
* Suspected peritoneal factor infertility
* Tubal or male factor infertility or sub-fertility

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | one year

SECONDARY OUTCOMES:
Ovulation rate Abortion rate Live-birth rate Adverse events | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Magna Graecia" of Catanzaro; Francesco Orio, MD, Principal Investigator — Department of Endocrinology, University "Federico II" of Naples; Achille Tolino, MD, Principal Investigator — Department of Obstetrics & Gynecology, University "Federico II" of Naples
Locations (1):
- Pugliese Hospital, Catanzaro, Catanzaro, CZ, Italy

REFERENCES:
- [Background] Palomba S, Orio F Jr, Falbo A, Russo T, Tolino A, Zullo F. Clomiphene citrate versus metformin as first-line approach for the treatment of anovulation in infertile patients with polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Sep;92(9):3498-503. doi: 10.1210/jc.2007-1009. Epub 2007 Jun 26. PMID 17595241
- [Background] Palomba S, Orio F Jr, Falbo A, Manguso F, Russo T, Cascella T, Tolino A, Carmina E, Colao A, Zullo F. Prospective parallel randomized, double-blind, double-dummy controlled clinical trial comparing clomiphene citrate and metformin as the first-line treatment for ovulation induction in nonobese anovulatory women with polycystic ovary syndrome. J Clin Endocrinol Metab. 2005 Jul;90(7):4068-74. doi: 10.1210/jc.2005-0110. Epub 2005 Apr 19. PMID 15840746
- [Background] Palomba S, Falbo A, Orio F Jr, Manguso F, Russo T, Tolino A, Annamaria C, Dale B, Zullo F. A randomized controlled trial evaluating metformin pre-treatment and co-administration in non-obese insulin-resistant women with polycystic ovary syndrome treated with controlled ovarian stimulation plus timed intercourse or intrauterine insemination. Hum Reprod. 2005 Oct;20(10):2879-86. doi: 10.1093/humrep/dei130. Epub 2005 Jun 15. PMID 15958399